CLINICAL TRIAL: NCT00144391
Title: Physiologic Testosterone Replacement in Women With Hypopituitarism
Brief Title: Testosterone Gel Applied to Women With Pituitary Gland Problems
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Theodore Friedman, Professor, Charles Drew University of Medicine and Science
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-02-511-07; 1U54HD041748-01 (NIH)
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-04

CONDITIONS: Panhypopituitarism
MeSH Terms: conditions — Combined Pituitary Hormone Deficiency

STUDY DESIGN:
Intervention Model Description: Testosterone and Placebo
Who Masked: Participant, Investigator
Masking Description: Testosterone and Placebo
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transdermal Testosterone Gel (Experimental): Transdermal Testosterone Gel (2 mg per pump), 2 pumps per day for 6 months
  Interventions: Drug: Transdermal Testosterone gel
- Placebo (Placebo Comparator): Placebo 2 pumps per day for 6 months
  Interventions: Drug: Transdermal Testosterone gel

INTERVENTIONS:
Drug: Transdermal Testosterone gel — 2.0 mg per pump of transdermal testosterone gel. Study patients receive either 2 pumps of transdermal testosterone gel per thigh per day or they receive 2 pumps per placebo gel per thigh per day for 6 months.

SUMMARY:
The principal aim of this study is to evaluate if application of testosterone gel leads to improvement in measures of sexual function, thinking ability and quality of life in women with dysfunction of the pituitary gland. A secondary purpose is to determine the effects of testosterone replacement on body composition and muscle function and strength.

DETAILED DESCRIPTION:
Testosterone is the principal male sex hormone but is also present in smaller amounts in women and may be important for their health. Among its likely actions in women are the building of bone and muscle mass, increase in interest in sex (libido) and effects on the mood. Testosterone is commercially available as a hormone replacement therapy for males with an absence or lack of testosterone production. Testosterone for males is mainly given in the form of shots or skin patches which have certain disadvantages such as pain from shots and skin rashes from patches. It is anticipated that this experimental gel application will produce levels of the drug in the normal range in women.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18-55
* Hypopituitarism with central adrenal and/or gonadal deficiencies. To qualify patients will need to have either 1 or 2 and they need to have 3:

  1. To diagnose central adrenal deficiency, patients not on glucocorticoid replacement will have an insulin tolerance test (ITT) (patients with cardiovascular disease will be excluded) in which 0.1U/kg of insulin will be given by iv and a peak cortisol value of less than 20ug/dl, associated with a glucose level of less than 40mg/dL will be considered consistent with central adrenal insufficiency. Patients on glucocorticoid replacement will be evaluated by examining their prior workup and if it is determined that they had evidence of central adrenal deficiency, an ITT will not be required to document central adrenal deficiency (an ITT will still be performed to determine GH deficiency).
  2. To diagnose central gonadal deficiency, patients will be asked if they had amenorrhea or oligomenorrhea prior to estrogen replacement. An FAH of less than 5 MIU/ML will be used to confirm that they have central and not primary gonadal deficiency. In select patients in which the diagnosis of central gonadal deficiency is unclear, we may perform an LHRH stimulation test, in which 100 ug iv of LHRH (Factrel) will be given and a peak LH response of less than 15 MIU/ML will be considered consistent with central gonadotropin insufficiency.
  3. Serum testosterone level on transdermal estrogen replacement of less than 20 ng/dL or free testosterone of less than 1.5 pg/ml.
* No other significant medical condition
* Weight between 80 and 150% of ideal body weight
* Able to provide informed consent
* All races and ethnicities
* All patients regardless of marital status and relationship status.

Exclusion Criteria:

* Physical disabilities that would prevent them from participating in the study.
* Current use of testosterone or other androgenic steroids. Patients who are taking testosterone, DHEA or other androgen precursors will discontinue these medications/supplements three months prior to the study.
* Significant cardiopulmonary disease (prior myocardial infarction causing ventricular dysfunction, angina, arrhythmias, congestive heart failure, valvular problem), venous thrombotic event (pulmonary embolism or deep vein thrombosis), renal disease (creatinine greater than 1.5 mg/dL), diabetes mellitus on insulin, uncontrolled hypertension, malignancy (other than basal cell skin carcinoma) or major psychiatric disease. Patients with depression or anxiety on a stable dose of medication will be allowed to enroll.
* Current abuse of illicit drugs or heavy ethanol use.
* History of breast cancer or abnormal mammogram at entry. If patients with an abnormal mammogram or PAP smear are appropriately evaluated and found not to have cancer, they will be allowed to participate in the study.
* Those with significant liver function abnormalities defined as SGOT, SGPT or alkaline phosphatase value of greater than one and one-half the upper limit of normal in our Clinical Pathology Laboratory or serum bilirubin levels of greater than 2 mg/dL will be excluded.
* Those with history of hyperandrogenic disorders such as hirsutism and polycystic ovary disease will be excluded. These conditions are rare in women with hypopituitarism. Testosterone administration to these patients may exacerbate the underlying disorder.
* Women who are pregnant, seeking to become pregnant in the next 6 months, or breast-feeding.
* Those who have previously experienced intolerance to other transdermal systems or gels
* Drugs known to alter testosterone production such as megace or ketoconazole.
* Patients with untreated hyperprolactinemia or active Cushing's disease. Patients with treated prolactinoma or Cushing's disease will be allowed to participate in the study.
* Hematocrit of greater than 50%
* Male sex
* Not willing to answer all questions on surveys
* EKG showing ischemia or prior myocardial infarction
* Patients with extensive brain surgery, severe head injury, brain tumors or other conditions that profoundly affect CNS function.
* Patients not willing to be placed on a standardized hormonal replacement regimen including transdermal estrogen and growth hormone.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2003-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore C Friedman, M.D., Ph.D., Principal Investigator — Charles Drew University of Medicine and Science
Locations (1):
- Charles Drew University of Medicine and Science, Los Angeles, California, United States

REFERENCES:
- See also: Clinical Trial Research site — http://www.centerwatch.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Transdermal Testosterone Gel: Transdermal Testosterone gel- 2.0 mg per pump dose 2 pumps per thigh per day for 6 months
- Placebo: Placebo
  placebo gel- 2 pumps per thigh per day for 6 months
Period: Overall Study
Arm/Group | Transdermal Testosterone Gel | Placebo
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Transdermal Testosterone Gel: 2.0 mg per pump dose. Study patients receive either 2 pumps per thigh per day of transdermal testosterone gel or 2 pumps of placebo per thigh per day for 6 months
  Transdermal Testosterone gel: 2.0 mg per pump of transdermal testosterone gel. Study patients receive either 2 pumps of transdermal testosterone gel per thigh per day or they receive 2 pumps per placebo gel per thigh per day for 6 months.
- Placebo: Placebo
  Transdermal Testosterone gel: 2.0 mg per pump of transdermal testosterone gel. Study patients receive either 2 pumps of transdermal testosterone gel per thigh per day or they receive 2 pumps per placebo gel per thigh per day for 6 months.
- Total: Total of all reporting groups
Arm/Group | Transdermal Testosterone Gel | Placebo | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (9) | 42 (14) | 43 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Fatigue Impact Scale
Description: change in fatigue impact scale there are 42 questions. Each question can be answered from 0 (no problem) to 4 (extreme problem), so a higher score indicates more severe fatigue impact. minimum score=0, maximum score =148 values are calculated at baseline and 6 months and the score at 6 months compared to baseline months is calculated
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transdermal Testosterone Gel | Placebo
Number analyzed (Participants) | 11 | 9
units on a scale | -22.9 (29.5) | 2.2 (30.7)
Statistical Analysis 1: Comparison: Transdermal Testosterone Gel vs Placebo; Test type: Superiority; p = 0.08, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Transdermal Testosterone Gel | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 1/11 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transdermal Testosterone Gel (N=11) | Placebo (N=9)
hirsutism (Endocrine disorders) | 1 (1) | 0 (0) — patient developed increase in facial hair, oily hair and acne

LIMITATIONS AND CAVEATS:
Small number of patients recruited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes